CLINICAL TRIAL: NCT06967389
Title: Mitigation of Cardiovascular Disease Risks in Children With Extreme Obesity (MODERN)
Brief Title: Mitigation of Cardiovascular Disease Risks in Children With Extreme Obesity
Acronym: MODERN
Status: Recruiting | Type: Observational
Sponsor: John Bauer (Other)
Responsible Party: Sponsor-Investigator, John Bauer, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: 98420
Record Dates: First submitted 2025-02-25; First posted 2025-05-13 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Obesity and Overweight; Obese Adolescents; Weight Management; Weight Loss; Cardiovascular Disease Risk Factor
Keywords: semaglutide; Wegovy; Ozempic; obesity; overweight; adolescent; weight management; weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss | interventions — semaglutide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine samples will be stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment Group: All participants in this study will be given the study drug.
  Interventions: Drug: Ozempic®

INTERVENTIONS:
Drug: Ozempic® — The study medication will be given in accordance with standard of care dosing schedule.

SUMMARY:
The goal of this clinical trial is to learn if the drug semaglutide changes markers of disease risk as it relates to weight in children ages 12-15 years old who are obese (class 2 or 3). The main questions it aims to answer are:

* How do the rate of weight loss, body mass index (BMI), body composition, heart structure and function, and exercise ability interact with one another in the study population at enrollment?
* How do risk markers of disease change over the study in the study participants who are given semaglutides to help with weight loss?
* Are there differences in the above factors between males and females and are there key factors to help improve the outcomes?

Participants will be given semaglutide for this study. During the course of the study, participants will:

* have two cardiac MRI scans OR two cardiac echocardiograms (one before starting semaglutide and one around 12 months after taking the drug)
* have body composition and fitness levels assessed twice (before semaglutide and around 12 months after taking it) and have urine specific gravity (USG) measured
* have extra blood drawn when labs their doctor orders are already being drawn (once at the beginning of the study, once around 6 months after enrollment, and once at the end of the study)
* have follow up visits with the study doctor
* be asked to take a pregnancy test if they are female and have started menstruation

DETAILED DESCRIPTION:
This is an observational study in which all participants will be given semaglutide. There will be no randomization and no placebo.

Participants will be in the study for 12 months (+/- 2 months) depending on when they reach the maintenance dose of semaglutide.

Blood and urine will be maintained by the principal investigator indefinitely. Identifiers will be removed from the samples.

Approximately 50 patients will be enrolled.

The study drug, Ozempic, is FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen at University of Kentucky Pediatric High BMI Clinic
* Diagnosis of Obesity Class 2 or 3
* Meeting the clinical criteria for the medical intervention with semaglutide for weight loss

Exclusion Criteria:

* Any current prescribed anti-obesity medications (AOM) such as Orlistat, Phentermine, Qsymia (Phentermine/Topiramate), Liraglutide, Semaglutide, and Setmelanotide
* Any current prescribed anti-hypertensive medications
* Any specific end-organ acute concerns (kidney disease, liver disease, congenital disease).
* Any active infections at enrollment.
* Any systemic steroid use longer than 3 month use or within the last month before enrollment (not including inhaled, ophthalmic, intranasal, and topical).
* Any limitations that would make exercise testing not possible.
* Any congenital abnormality or genetic syndrome known to be associated with obesity
* Pregnancy
* Inability to receive an MRI
* Personal or family history of medullary thyroid carcinoma (per product insert)
* Patients with Multiple Endocrine Neoplasia syndrome type 2 (per product insert)

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited from the University of Kentucky's High BMI and/or Pediatric Nephrology Clinics.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in medication use | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  This will be assessed by reviewing changes in the electronic medical record
Change in Lipid Profile | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  plasma/serum samples will be analyzed. blood lipid panel to include total cholesterol (mg/dL), HDL (mg/dL), triglycerides (mg/dL), and LDL (mg/dL) will be assessed
Change in C-reactive protein | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  data obtained from blood samples
Change in Tumor necrosis factor | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  data obtained from blood samples
Change in Interleukin-6 | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  data obtained from blood samples
Change in Adiponectin | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  data obtained from blood samples
Change in Soluble Intercellular Adhesion Marker | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  data obtained from blood samples
Changes in Renin-Angiontensin-Alsosterone System biomarkers profiling | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Changes in RAAS biomarkers at the defined study points will be evaluated.
Change in Systolic Blood pressure | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
Change in Diastolic Blood pressure | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Blood pressure (systolic/diastolic) (mmHg) ambulatory blood pressure monitoring (ABPM) (mmHg) will be taken at the listed timepoints.
Change in ambulatory blood pressure | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
Change in Cardiac structure | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Changes from baseline cardiac MRI and/or cardiac echocardiograms (ECHO) will be assessed including overall heart and chamber size, wall thickness, etc.
Change in Cardiac function (Ejection Fraction) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Changes from baseline cardiac MRI and/or cardiac echocardiograms (ECHO) will be assessed.
Change in Cardiac function (Stroke Volume (SV) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Changes from baseline cardiac MRI and/or cardiac echocardiograms (ECHO) will be assessed.
Change in Cardiac function (Cardiac Output (CO) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Changes from baseline cardiac MRI and/or cardiac echocardiograms (ECHO) will be assessed.
Change in Cardiac function (Wall motion) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Changes from baseline cardiac MRI and/or cardiac echocardiograms (ECHO) will be assessed.
Change in Cardiac function (Valve motion) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Changes from baseline cardiac MRI and/or cardiac echocardiograms (ECHO) will be assessed.

SECONDARY OUTCOMES:
Change in Dietary habits | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  It assesses the frequency and quality of dietary habits, such as the consumption of fruits, vegetables, whole grains, and unhealthy foods like sugary snacks and fast food.
  The scoring is typically based on a scale representing frequency:
  0 = Never or less than once per week, 1 = 1-2 times per week, 2 = 3-4 times per week, 3 = 5-6 times per week, 4 = Daily or more.
  Higher scores on the healthy scale = better dietary habits
Change in exercise habits | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Assessed with the BMI Clinic dietary and exercise habit survey in which participants record the frequency of activities.
  It assesses the frequency, duration, and/or intensity of physical activity (e.g., walking, moderate activity, vigorous activity, including aerobic and strength training).
  For interpretation:
  High Score: Indicates sufficient physical activity Low Score: Suggests insufficient physical activity
Patient Health Questionnaire-9 (PHQ-9) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  The PHQ-9 is a 9-item self-report questionnaire that is widely used to assess depression symptom severity. A PHQ-9 score ≥10 has a sensitivity of 88% and a specificity of 88% for major depression. PHQ-9 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe depression, respectively. Higher scores indicating greater depression severity.
Generalized Anxiety Disorder-7 questionnaire (GAD-7) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  A 7 item self-complete questionnaire with very good sensitivity (89%) and specificity (82%) for Generalised Anxiety Disorder (GAD). Response scores for each item ranging from 0 (not at all) to 3 (every day). The range for the total score is 0 to 21, with higher scores representing greater symptoms of anxiety
Change in Anthropomorphic outcomes - Body Mass Index (BMI) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
Change in Anthropomorphic outcomes - Waist circumference | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
Change in Anthropomorphic outcomes - Bioimpedence | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Whole-body electrical resistance will be measured with the subjects using the BodyStat Quadscan 4000 Bioelectric Impedance Analyzer
Change in Anthropomorphic outcomes - Resting metabolic rate | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  A handheld resting metabolic rate (RMR) calculator/indirect calorimeter (MedGem RMR) will be used to estimate the RMR (caloric needs).
Change in Anthropomorphic outcomes - Cardiorespiratory Fitness | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  Maximal Graded Exercise Testing (Maximal GXT): The maximal graded exercise tests will be performed using an indirect calorimetry testing system
Change in complete blood count (CBC) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  plasma/serum samples will be analyzed
Change in Liver panel profile | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  -plasma/serum samples will be analyzed. The individual components are grouped as a panel to for an overall evaluation of the system's functioning
Change in Renal panel profile | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  -plasma/serum samples will be analyzed. The individual components are grouped as a panel to for an overall evaluation of the system's functioning
Change in Thyroid panel profile | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  -plasma/serum samples will be analyzed. The individual components are grouped as a panel to for an overall evaluation of the system's functioning
Change in Fasting glucose | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  -plasma/serum samples will be analyzed
Change in Fasting Insulin | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment
  -plasma/serum samples will be analyzed
Change in hyperglycemia assessed by Homeostatic Model Assessment of Insulin Resistance, (HOMA-IR) | Enrollment, 6 months post enrollment, 12 months +/- 2 months post enrollment

CONTACTS AND LOCATIONS:
Overall Officials: John Bauer, PhD, Study Chair — University of Kentucky; Margaret Murphy, RD PhD, Principal Investigator — University of Kentucky; Aurelia Radulescu, MD, Study Director — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes